CLINICAL TRIAL: NCT06118008
Title: A Multiple-dose, Randomized, Double-blind, Placebo and Positive Controlled Phase IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HS-20094 in Subjects With Type 2 Diabetes.
Brief Title: A Study of HS-20094 in T2DM Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-20094-201
Record Dates: First submitted 2023-05-25; First posted 2023-11-07 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- HS-20094 5mg (Experimental): Drug: HS-20094 Administrated by subcutaneous injection
  Drug: Placebo Administrated by subcutaneous injection
  Drug: Semaglutide Administrated by subcutaneous injection
  Interventions: Drug: HS-20094 5mg
- HS-20094 10mg (Experimental): Drug: HS-20094 Administrated by subcutaneous injection
  Drug: Placebo Administrated by subcutaneous injection
  Drug: Semaglutide Administrated by subcutaneous injection
  Interventions: Drug: HS-20094 10mg
- HS-20094 15mg (Experimental): Drug: HS-20094 Administrated by subcutaneous injection
  Drug: Placebo Administrated by subcutaneous injection
  Drug: Semaglutide Administrated by subcutaneous injection
  Interventions: Drug: HS-20094 15mg
- HS-20094 20mg (Experimental): Drug: HS-20094 Administrated by subcutaneous injection
  Drug: Placebo Administrated by subcutaneous injection
  Drug: Semaglutide Administrated by subcutaneous injection
  Interventions: Drug: HS-20094 20mg

INTERVENTIONS:
Drug: HS-20094 5mg — Administrated by subcutaneous injection
  Other Names: HS-20094 injection 5mg
  Arms: HS-20094 5mg
Drug: HS-20094 10mg — Administrated by subcutaneous injection
  Other Names: HS-20094 injection 10mg
  Arms: HS-20094 10mg
Drug: HS-20094 15mg — Administrated by subcutaneous injection
  Other Names: HS-20094 injection 15mg
  Arms: HS-20094 15mg
Drug: HS-20094 20mg — Administrated by subcutaneous injection
  Other Names: HS-20094 injection 20mg
  Arms: HS-20094 20mg

SUMMARY:
This is a randomized, placebo and active-control, multiple-dose, phase IIa trial. Patients were randomly assigned to receive HS-20094 (12 patients), placebo (3 patients), or active control drug Semaglutide injection (3 patients) in a 4:1:1 ratio to each of four dose cohorts of 5 mg, 10 mg, 15 mg, and 20 mg. HS-20094 and placebo were administered in a double-blind design by subcutaneous injection once a week for a total of four times, and the dose was gradually increased weekly (2.5-2.5-5-5 mg, 5-510-10 mg, 5-10-15-15 mg, 5-10-15-20 mg). The active control drug semaglutide was administered by open-label, titrated subcutaneous injection once a week for a total of four times, and the dose was increased gradually every week until 1.0 mg (0.25-0.5-0.5-1.0 mg). The primary study objective was to 1) Evaluate the safety and tolerability of multiple subcutaneous injections of HS-20094 in subjects with type 2 diabetes mellitus (T2DM) with or without overweight or obesity;2) Evaluate the pharmacokinetics, pharmacodynamics and immunogenicity of multiple subcutaneous injections of HS-20094.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects,20-65 years of age at the time of signing informed consent.
* Type 2 diabetes mellitus diagnosed for at least 3 months before the screening visit.
* Treated with conventional lifestyle intervention and stable treatment with metformin ( ≥ 1000 mg/day) at least 3 months prior to screening HbA1c 7.5-10%(both inclusive)at screening visit.

Exclusion Criteria:

* A history of type 1 diabetes, specific diabetes, or secondary diabetes.
* Presence of-clinically significant lab or ECG results that may affect the evaluation of the efficacy or safety of the study drug at screening visit.
* Acute or chronic pancreatitis at any time before screening, or serum lipase/amylase above the upper limit of normal at screening.
* A history of grade 2 hypoglycemia(blood glucose 3.0 mmol/L)or grade 3 hypoglycemia(hypoglycemia with a serious event of consciousness and/or physical alteration requiring assistance from another person for recovery)within 6 months before screening.
* Diabetid ketoacidosis or hyperosmolar coma or lactic acidosis requiring hospitalization occurred within 6 months before screening.
* Severe infection such as diabetic foot infection, pneumonia, or sepsis within 30 days before screening.
* Uncontrollable hypertension.
* History of acute cardiovascular and cerebrovascular diseases within 6 months prior to screening.
* Any organ-system malignancies developed within 5 years except for cured local basal cell carcinoma of the skin and carcinoma in situ of the cervix.
* Pregnant or lactating woman.
* In the investigator's judgment, there were circumstances that affected subject safety or otherwise interfered with the evaluation of results.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse event (AE), serious adverse event (SAE), AE leading to study discontinuation, AE severity and relation with study drug | From Baseline to Day 57.
  A summary of AEs and SAEs, AE leading to study discontinuation, AE severity and relation with study drug will be reported in the reported adverse events module
The number of participants with changes of laboratory tests blood routine, urine routine, blood biochemistry, coagulation function | From Baseline to Day 57
The changes ECG examination assessed by PR, R-R, QRS and QTcF | From Baseline to Day 57
  12-lead electrocardiogram (ECG) parameters
The changes in Blood pressure | From Baseline to Day 57
  Vital signs
Pulse rate | From Baseline to Day 57
  Vital signs
Respiratory rate | From Baseline to Day 57
  Vital signs
Temperature | From Baseline to Day 57
  Vital signs

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Cmax of HS-20094 | Baseline to Day 57
  PK: Cmax of HS-20094
Pharmacokinetics (PK): Tmax of HS-20094 | Baseline to Day 57
  PK: Tmax of HS-20094
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of HS-20094 | Baseline to Day 57
  PK: AUC of HS-20094
Pharmacodynamics (PD): HbA1c | Baseline to Day 29
  PD: change of HbA1c

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No